CLINICAL TRIAL: NCT01742949
Title: Evaluation of Advantages Linked to the Use of Humidification by ThermoSmart During Continuous Positive Airway Pressure
Brief Title: Study to Predict the Benefits of First-line Humidification Use and Comparison of the Effect of ThermoSmart™ and no Humidification on Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FPH-TS2012
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thermosmart (Active Comparator): Subjects receive heated humidification
  Interventions: Device: Heated humidification (ThermoSmart)
- No humidification (Placebo Comparator): Subjects use dry CPAP / APAP
  Interventions: Device: No Humidification

INTERVENTIONS:
Device: Heated humidification (ThermoSmart) — Heated Humidification (ThermoSmart) Turned On
  Arms: Thermosmart
Device: No Humidification — Heated Humidification (ThermoSmart) Turn Off
  Arms: No humidification

SUMMARY:
This study aims to investigate the benefits of using first line heated humidification. The primary objective of this research is to determine the effect of high levels of humidification delivered by ThermoSmart™ on CPAP adherence. In addition, to determine if it is possible to predict which patients benefit the most (i.e. be more adherent with therapy) from high levels of humidification delivered by ThermoSmart.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Diagnosed with OSA and eligible for CPAP treatment under local requirements (AHI>30 or if AHI is lower than 30, at least 10 micro arousals identified during diagnosis PSG).
* Naïve to CPAP therapy, i.e have not been prescribed, or used CPAP in the last 5 years
* Patients receiving social security coverage (excluding MEAs)
* Fluent spoken and written French

Exclusion Criteria:

* Severe heart disease
* Co-existing lung disease
* Co-existing sleep disorder
* Pregnant
* Refused participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pia D'Dortho, MD, Principal Investigator — Hôpital Bichat-Claude Bernard
Locations (4):
- France (4):
  - Hôpital Bichat-Claude Bernard, Paris, Paris Cedex
  - Hôpital Henri Mondor, Paris
  - Hôpital La Pitie Salpetriere, Paris
  - Hôpital Louis Mourier, Paris

RESULTS

PARTICIPANT FLOW:
Groups:
- Thermosmart On, Then Followed by ThermoSmart Off: Subjects receive heated humidification (ThermoSmart) first, then followed by it off.
- ThermoSmart Off, Then Followed by ThermoSmart On: Subjects receive dry CPAP/APAP (no ThermoSmart), then followed by it on.
Period: Overall Study
Arm/Group | Thermosmart On, Then Followed by ThermoSmart Off | ThermoSmart Off, Then Followed by ThermoSmart On
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Participants as this is a crossover trial where participant will experience both heated humidification (ThermoSmart On) or dry CPAP/APAP (ThermoSmart Off)
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.379)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Adherence with treatment per night averaged over total time period measured via internal software on the CPAP device and reported using InfoSmart™ software. The report will include all the supporting information recorded within the CPAP device.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Thermosmart | No Humidification
Number analyzed (Participants) | 40 | 40
hours per night | 4.7 (2.7) | 5.0 (2.5)

2. Secondary Outcome: Epworth Sleepiness Score
Description: Subjective measure of daytime sleepiness. There are 8 questions where the patient picks a scale of 0 = would never doze to 3 = high level of dozing for each questions. There can be a total score of 24. A score of 0-10 indicates normal daytime sleepiness, 11-12 mild excessive daytime sleepiness, 13-15 moderate excessive daytime sleepiness and 16-24 is severe excessive daytime sleepiness.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thermosmart | No Humidification
Number analyzed (Participants) | 40 | 40
units on a scale | 6.2 (0.8) | 6.0 (0.6)

3. Secondary Outcome: Short Functional Outcomes of Sleep Questionnaire (FOSQ-10)
Description: Collected through the Short Functional Outcomes of Sleep Questionnaire (FOSQ-10). The questionnaire has 10 questions which ask how daytime sleepiness has impacted their quality of life. Each question has a scale of 1 = yes extreme to 4 = No. Lower total score (min 10) means that the disease is affecting your quality of life while a higher total score (maximum 40) means that the disease is not affecting your quality of life.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thermosmart | No Humidification
Number analyzed (Participants) | 40 | 40
units on a scale | 32.1 (5.6) | 32 (6.2)

4. Secondary Outcome: Subjective Dry Nose
Description: Measured through a visual analog scale. The patient has to mark a cross on the scale to indicate the severity of their symptoms. On the left side of the scale has "not at all" and on the right side of the scale has "extremely", In order to analyze the data, a ruler from the start of the scale (Left side) to the middle of the cross is measured in cm. The total length of the scale is 14 cm. Therefore, the minimum score is 0 and the maximum score is 14. The higher the score means that the participant is experiencing more symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thermosmart | No Humidification
Number analyzed (Participants) | 40 | 40
units on a scale | 3.1 (3.6) | 4.8 (4.9)

5. Secondary Outcome: Subjective Dry Mouth
Description: as for outcome 4
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thermosmart | No Humidification
Number analyzed (Participants) | 40 | 40
units on a scale | 5.2 (4.9) | 6.7 (4.9)

6. Secondary Outcome: Subjective Sinusitis
Description: as for outcome 4
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thermosmart | No Humidification
Number analyzed (Participants) | 40 | 40
units on a scale | 1.8 (2.7) | 2.5 (3.6)

7. Secondary Outcome: Preference
Description: Through a questionnaire, the participant is asked to picked rather they prefer treatment A (No ThermoSmart) or treatment B (ThermoSmart). If they did not pick neither, it is considered no preference.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Thermosmart: Subjects preferring ThermoSmart
- No Humidification: Subjects preferring No ThermoSmart
- No Preference: No Preference for ThermoSmart or no ThermoSmart
Arm/Group | Thermosmart | No Humidification | No Preference
Number analyzed (Participants) | 40 | 40 | 40
Participants | 26 | 11 | 3

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Thermosmart | No Humidification
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No